CLINICAL TRIAL: NCT06597708
Title: Dietary Diversities: Exploring the Influence of Keto Diet and Intermittent Fasting on Oral Health and Salivary Inflammatory Biomarkers
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Al-Mustansiriyah University (Other)
Responsible Party: Principal Investigator, Sarah Thamer Kadhum, Dentist, Al-Mustansiriyah University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: MUPRV010
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Gingivitis
MeSH Terms: conditions — Gingivitis | interventions — Diet, Ketogenic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- participants committed to keto diet (Active Comparator): The experimental intervention consisted of a KD without caloric restriction over a period of 4 weeks. Prior to the study period, the participants were instructed by a dietitian. The participants were provided with online brochure describing the main aspects of a KD and given a list of suitable foods with a very low carbohydrate content. They were advised to eat ad libitum but to limit their carbohydrate intake to a maximum of 20-40 g/day to derive at leasut 75%, 15-20%, and 5-10% of total energy from fats, protein, and carbohydrates, respectively. The participants were allowed to vary the food according to their preferences within the framework of the KD.
  Interventions: Behavioral: keto diet
- participants committed to intermittent fasting with calorie restriction (Active Comparator): The 16/8 TRF group was asked to consume their daily calorie intake during an 8-hour window during the daytime and then fast for the remaining 16 hours each day throughout the intervention period. During the 16 hours fasting, they were able to drink water, coffee and tea without sugar. Participants are encouraged to drink 6-8 glasses of water per day. They were free to arrange the 8-hour eating window based on personal preferences. This flexibility was expected to help the participants adapt to their individual lifestyles and to facilitate compliance with the dietary intervention.
  Interventions: Behavioral: intermittent fasting with calorie restriction

INTERVENTIONS:
Behavioral: keto diet — They were advised to eat ad libitum but to limit their carbohydrate intake to a maximum of 20-40 g/day to derive at leasut 75%, 15-20%, and 5-10% of total energy from fats, protein, and carbohydrates, respectively.
  Arms: participants committed to keto diet
Behavioral: intermittent fasting with calorie restriction — The 16/8 TRF group was asked to consume their daily calorie intake during an 8-hour window during the daytime and then fast for the remaining 16 hours each day throughout the intervention period.
  Arms: participants committed to intermittent fasting with calorie restriction

SUMMARY:
This study aims to investigate the impact of short term, two distinct dietary interventions, namely the Keto diet and Intermittent Fasting on oral health by measuring the severity of:

* Periodontal diseases (Gingivitis).
* Oral health status (Plaque index). As well as measuring the impact of these different dietary pattern on the levels of C- Reactive Protein, IL-6, TNF-a in mean of inflammatory biomarkers as well as LL- 37 peptide as well as measuring salivary flow and ph.

Objectives of the study

1. Evaluate the impact of Keto diet and Intermittent Fasting on oral health among the Iraqi population.
2. Assess changes in inflammatory biomarkers within the study groups before and after the intervention period.
3. Compare the effects of Keto diet and Intermittent Fasting on oral health and inflammatory biomarkers between the two intervention groups.
4. Examine the variations in oral health and inflammatory biomarkers within each group by comparing the baseline (Iraqi diet) and post-intervention stages.
5. Investigate the influence of Keto diet and Intermittent Fasting on the levels of LL37, an antimicrobial peptide.

ELIGIBILITY:
Inclusion Criteria:

* Adults in good general health with a BMI in the range of 19-30 kg/m2 (overweight and obese cl I).
* Age 20-35 years.

Exclusion Criteria:

* low-carbohydrate nutrition already prior to the study.
* Impaired liver and renal function, kidney stones.
* Pregnancy or lactation period
* Diabetes mellitus and any fatty acid-metabolism disorders.
* Presence of systemic disease (diabetes, hypertension, cardiovascular disease) that may affect oral health.
* Medications that may affect periodontal health conditions.
* Use of anti-inflammatory and antibiotic drugs during the last month before the examination.
* Smoking.
* Use of dietary supplements.
* Wearing orthodontics or prosthodontics appliances.

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
effect of keto diet on oral health | 30 days
  effect of keto diet on oral health by measuring the plaque index and bleeding on probing index
effect of intermittent fasting on oral health | 30 days
  effect of intermittent fasting on oral health by measuring the plaque index and bleeding on probing index

SECONDARY OUTCOMES:
The effect of keto diet on salivary inflammatory biomarkers | 30 days
  effect of keto diet on salivary inflammatory biomarkers ( IL-6, IL-1B, C-RP, TNF-A, LL-37)
The effect of intermittent fasting on salivary inflammatory biomarkers | 30 days
  effect of intermittent fasting on salivary inflammatory biomarkers ( IL-6, IL-1B, C-RP, TNF-A, LL-37)
comparing the effect of KD and IF on inflammatory biomarkers | 30 days
  comparing the effect of keto diet and intermittent fasting on salivary inflammatory biomarkers ( IL-6, IL-1B, C-RP, TNF-A, LL-37)
comparing the effect of KD and IF on oral health | 30 days
  comparing the effect of KD and IF on oral health by measuring the plaque index and bleeding on probing index
The effect of intermittent fasting on bodyweight | 30 days
  The effect of intermittent fasting on bodyweight loss for overweight and obese cl I participants
The effect of keto diet on bodyweight loss | 30 days
  The effect of keto diet on bodyweight loss for overweight and obese cl I participants
The effect of keto diet on salivary PH | 30 days
  The effect of keto diet on salivary PH ( an increase or decrease)
The effect of intermittent fasting on salivary PH | 30 days
  The effect of intermittent fasting on salivary PH ( an increase or decrease)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Mustansiriyah, Baghdad, Street 6, Iraq